CLINICAL TRIAL: NCT07135687
Title: Oral Losartan to Decrease the Risk of Postoperative Arthrofibrosis Following Primary and Revision Anterior Cruciate Ligament Reconstruction
Brief Title: Study to Use Oral Losartan to Decrease the Risk of Postoperative Scarring Following (ACL) Reconstruction
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: Arthroscopy Association of North America (AANA) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 24120601
Record Dates: First submitted 2025-08-14; First posted 2025-08-22 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: ACL Injury; ACL Reconstruction; Scar Formation
Keywords: ACL; Postoperative Arthrofibrosis; Losartan
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — Losartan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Losartan (Experimental): The experimental arm (Arm 1) will receive 25mg losartan daily for 3 days followed by 50 mg losartan daily for 25 days.
  Interventions: Drug: Losartan
- Placebo (Placebo Comparator): The placebo arm (Arm 2) will receive a placebo tablet with the same appearance and frequency to that of the losartan group.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Losartan — Two types of losartan capsules will be compounded by combining a broken-up 25mg or 50mg losartan tablet and microcrystalline cellulose placebo filler to eliminate rattling of the broken tablet inside of the capsule. The 25mg losartan capsules will be yellow and the 50 mg losartan capsules will be blue.
  Arms: Losartan
Other: Placebo — The placebo capsules will consist of microcrystal cellulose and will come in yellow and blue to appear identical to the losartan capsules.
  Arms: Placebo

SUMMARY:
The purpose of this study to investigate the effect of using losartan (a blood pressure lowering drug with anti-scarring properties) on preventing primary postoperative arthrofibrosis (formation of abnormal scar tissue) in the knees in participants undergoing anterior cruciate ligament (ACL) repair surgery of their knee.

DETAILED DESCRIPTION:
Losartan, an angiotensin-II receptor blocker (ARB), approved by the Food and Drug Administration (FDA) for the treatment of hypertension and diabetic nephropathy, has garnered recent interest in the field of orthopedic surgery as an anti-fibrotic (anti-scarring) agent. Losartan's primary mechanism of action as an anti-hypertensive involves acting as a receptor antagonist for angiotensin II, a peptide produced by the liver which causes vasoconstriction, release of anti-diuretic hormone from the pituitary gland, and release of aldosterone from the adrenal glands, among other functions. Losartan secondary function is to act as a TGF-β1 blocker. TGF-β1 has been implicated in pro-fibrotic pathways in multiple organs systems. Losartan, initially as a treatment for hypertension and diabetic nephropathy, was found to have benefits against fibrosis in the renal system. As a result, the use of losartan has gained interest in several other fields in medicine, including plastic surgery for wound healing and keloid prevention, in ophthalmology to prevent corneal scarring, and orthopedic surgery. The potential use of losartan presents an attractive anti-fibrotic prophylaxis candidate against the formation of postoperative arthrofibrosis following ACLR.

ELIGIBILITY:
Inclusion Criteria:

* Must be undergoing a primary ACLR with or without the following:
* Chondroplasty
* Synovectomy
* Loose body removal
* Removal of hardware
* Meniscal surgery (excluding meniscal allograft transplantation/MAT)
* Lateral extra-articular tenodesis
* Must have skeletal maturity in the distal femur and proximal tibial physes
* Must be age 18 years or older at time of enrollment

Exclusion Criteria:

* <18 years at time of enrollment
* No diagnosis of ACL tear
* ACL repairs
* Revision ACL reconstructions
* Open distal femur or proximal tibia physes
* Major concomitant procedures (such as osteotomy, MAT, or cartilage restoration surgery)
* History of prior proximal or distal femur fracture (including those receiving nonoperative treatment)
* History of prior ipsilateral femur or tibia osteomyelitis
* Medical history
* History of hypotensive disease, including postural orthostatic hypotension syndrome (POTS), autonomic dysreflexia, or Shy-Drager syndrome (aka multiple system atrophy), baseline hypotension <90 systolic or <60 diastolic mmHg.
* History of significant hepatic disease (liver transplantation, cirrhosis of any cause, or any liver disease with Child-Pugh classification B or C) due to hepatic metabolism of ARBs.
* Chronic kidney disease
* Rheumatologic disorders on immunologic medications
* Current medications including diuretics (i.e. furosemide), lithium, and spironolactone
* Current hypertension with prescription of an ARB or ACE-I
* Allergy to losartan
* Current pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2026-08 (Estimated); Primary Completion 2028-10 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Range of Motion | 12 months
  Range of motion measured from baseline to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Chahla, MD, PhD, Principal Investigator — Rush University Medical Center; Andrew Bi, MD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-08-13): https://cdn.clinicaltrials.gov/large-docs/87/NCT07135687/Prot_SAP_000.pdf